CLINICAL TRIAL: NCT00962039
Title: Anxiety and Recurrent Abdominal Pain in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: John V. Campo, M.D. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, John V. Campo, M.D., Chief Of Child & Adolescent Psychiatry -Medical Director, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5R01MH069715-04 (NIH); 5R01MH069715-04 (NIH); DAHBR B4-TBI
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Pain; Anxiety
Keywords: Abdominal Pain; Anxiety
MeSH Terms: conditions — Abdominal Pain; Anxiety Disorders | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Citalopram (Experimental): Citalopram was initiated at 10 mg daily for one week, with dosage increased to 20 mg daily during week 2, with an optional increase to 40 mg daily at week 4 or thereafter if response was judged to be suboptimal (CGI-I or CGI-S > 2).
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Placebo administered in capsules identical to those containing citalopram using microcrystalline cellulose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Participants will be randomly assigned to citalopram or placebo in a parallel groups design for 8 weeks of double-blind treatment beginning with 10 mg per day week 1, 20 mg per day week 2, and 40 mg per day week 4 or thereafter if response is suboptimal and there are no significant side effects.
  Other Names: Celexa
  Arms: Citalopram
Drug: Placebo — Participants will be randomly assigned to citalopram or placebo in a parallel groups design for 8 weeks of double-blind treatment beginning with 10 mg per day week 1, 20 mg per day week 2, and 40 mg per day week 4 or thereafter if response is suboptimal and there are no significant side effects.
  Arms: Placebo

SUMMARY:
This study aims to determine whether citalopram is a useful, well-tolerated, and safe treatment for children and adolescents ages 7 to 18 years with functional abdominal pain. The study hypothesis is that citalopram will be better than placebo in producing clinical improvement and reductions in abdominal pain. It is also hypothesized that citalopram and placebo will not differ in terms of safety and tolerability.

DETAILED DESCRIPTION:
This study aims to determine the relative efficacy, tolerability, and safety of the citalopram in the treatment of pediatric functional recurrent abdominal pain (FAP) in children and adolescents ages 7 to 18 years, inclusive. The goal is to recruit and randomize 100 subjects to citalopram or placebo. Secondary aims include to determine if citalopram is superior to placebo in reducing comorbid anxiety and depressive symptoms in children and adolescents with FAP, to explore potential mediators (i.e., anxiety, depression) and moderators (e.g., age, gender, referral from primary or specialty care) of treatment response, and to explore the durability and tolerability of citalopram treatment 18 weeks following completion of the double-blind treatment phase with the goal of generating data useful to the development of future studies. The study is novel in conducting recruitment, assessment, and treatment in traditional medical settings. Limited exclusion criteria and the delivery of study assessments and interventions within routine practice settings provide for considerably greater external validity than the typical efficacy study.

Study hypotheses:

1. Citalopram will be superior to placebo in producing clinical improvement and reductions in abdominal pain.
2. Citalopram and placebo will not differ in tolerability or safety.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 episodes of abdominal pain during the previous 3 months associated with functional impairment in the absence of explanatory physical disease following clinically appropriate medical assessment.
* Age 7 years 0 months to 18 years 11 months, inclusive, at initial evaluation.
* Significant global functional impairment as reflected by a score less than 70 on the Children's Global Assessment Scale
* Residing with a primary caretaker (i.e., parent, legal guardian, relative functioning as a parent, or foster parent) who has known the child well for at least 6 months prior to study entry and has legal authority to consent to participation.

Exclusion Criteria:

* Physical disease sufficient to explain the subjective distress and functional impairment suffered by the subject.
* FAP with atypical features:

  1. Abnormal abdominal or rectal examination
  2. GI bleeding (i.e., hematest positive stool or hematemesis)
  3. History of recurrent or persistent fever associated with the abdominal pain
  4. Involuntary weight loss (> 5% of body weight) over the previous 3 months
  5. Previous laboratory evidence suggesting explanatory physical disease
  6. Persistent nighttime awakenings due to abdominal pain (at least once per week and > 4 per month)
  7. Persistent or bilious vomiting (at least once per week and > 4 per month)
  8. Abdominal pain exclusively associated with menstruation
  9. Dysuria
* Physical disease in which citalopram monotherapy or study participation might prove to be disadvantageous or incompatible with quality care, including bleeding disorder characterized by prolonged bleeding time, uncontrolled epilepsy, or poorly controlled diabetes mellitus.
* Psychiatric problem or disorder in which citalopram monotherapy or study participation might prove to be disadvantageous or incompatible with quality care, including evidence that the child is a serious acute danger to self or others, anorexia nervosa, bulimia nervosa, schizophrenia, schizoaffective disorder, alcohol or substance abuse/dependence, or bipolar disorder.
* History of mental retardation as defined by full scale IQ < 70 on previous testing or participation in special education placement for mild to severe mental retardation.
* Inadequate English speaking abilities of child or parent(s) to complete study measures and/or communicate with study examiners.
* Adequate prior trial of citalopram, escitalopram, or another selective serotonin reuptake inhibitor or venlafaxine. Adequate trial is defined as at least 4 weeks of citalopram 20 mg/day, escitalopram 10 mg/day, fluoxetine 20 mg/day, fluvoxamine 100 mg/day, paroxetine 20 mg/day, sertraline 50 mg/day, or venlafaxine 75 mg/day.
* Concurrent use of non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, or anticoagulant medications.
* Treatment for physical or psychiatric illness initiated within the prior 4 weeks or escalating in dosage or intensity.
* History of hypersensitivity to citalopram or serotonin-syndrome.
* Participation in any investigational drug study within thirty days of study entry.
* Pregnancy
* Sexually active female subjects refusing to use a medically accepted method of birth control during the study, or who engaged in unprotected sexual activity during the 30 days prior to the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2004-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John V Campo, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campo JV, Perel J, Lucas A, Bridge J, Ehmann M, Kalas C, Monk K, Axelson D, Birmaher B, Ryan N, Di Lorenzo C, Brent DA. Citalopram treatment of pediatric recurrent abdominal pain and comorbid internalizing disorders: an exploratory study. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1234-42. doi: 10.1097/01.chi.0000136563.31709.b0. PMID 15381890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were clinically referred from primary care and specialty pediatric gastroenterology and were impaired as reflected by a score of less than 70 on the Children's Global Assessment Scale (CGAS).
Pre-assignment Details: Potential subjects with physical disease responsible for the abdominal pain, eating disorder, bipolar disorder, psychosis, alcohol/drug abuse, intellectual disability (IQ < 70), pregnancy, or prior trial of SSRI antidepressant or venlafaxine were excluded.
Groups:
- Citalopram: Citlaopram: Participants were randomly assigned to citalopram or placebo in a parallel groups design for 8 weeks of double-blind treatment beginning with 10 mg per day week 1, 20 mg per day week 2, and 40 mg per day week 4 or thereafter if response was suboptimal and there were no significant side effects.
- Placebo: Placebo: Participants were randomly assigned to citalopram or placebo in a parallel groups design for 8 weeks of double-blind treatment beginning with 10 mg per day week 1, 20 mg per day week 2, and 40 mg per day week 4 or thereafter if response was suboptimal and there were no significant side effects.
Period: Overall Study
Arm/Group | Citalopram | Placebo
Started | 40 | 41
Completed | 35 | 37
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Citalopram; Placebo: This double blind, placebo-controlled trial randomized 81 subjects ages 7 to 18 years in parallel groups to citalopram (n=40) or placebo (n=41) for 8 weeks. Citalopram was initiated at 10 mg per day week 1, 20 mg per day week 2, and 40 mg per day week 4 or thereafter if response was suboptimal and there were no significant side effects. Subjects were recruited by clinical referral from both the primary care and specialty pediatric gastroenterology clinical settings. In addition to meeting criteria for FAP, subjects were required to be significantly impaired as reflected by a score of less than 70 on the Children's Global Assessment Scale (CGAS). Potential subjects with physical disease responsible for the observed abdominal pain, eating disorder, bipolar disorder, psychosis, alcohol/drug abuse, intellectual disability (IQ < 70), pregnancy, or prior trial of SSRI antidepressant or venlafaxine were excluded.
- Total: Total of all reporting groups
Arm/Group | Citalopram | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 41 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale - Improvement (CGI-I) Will be Used to Assess Overall Global Illness Improvement. CGI-I Scores of 1 (Very Much Improved) or 2 (Much Improved) Indicate an Acceptable Treatment Response.
Description: Clinical Global Impression Scale - Improvement (CGI-I) is a 7-point scale, with lower values being more favorable, used to assess overall global illness improvement. The CGI is a clinician-completed measure, with values ranging from 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), to 7 (very much worse). CGI-I scores of 1 (very much improved) or 2 (much improved) were considered to indicate an acceptable treatment response. A global measure of functional status was chosen as a primary outcome due to the broad array of symptomatology seen in pediatric RAP and the ambiguous relationship between functional status and symptoms of pain, anxiety, and depression in pediatric RAP. The CGI-I is a dichotomous primary outcome measure of global clinical improvement with clinical response be defined as a CGI-I score of 1 or 2 for at least two consecutive weeks.
Time Frame: The CGI will be completed at weeks 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  CGI-I Week 2 | 3.48 [3.25 to 3.72] | 3.68 [3.44 to 3.93]
  CGI-I Week 4 | 3.03 [2.78 to 3.28] | 3.38 [3.09 to 3.67]
  CGI-I Week 8 | 2.65 [2.23 to 3.07] | 3.24 [2.88 to 3.61]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.92, Chi-squared — Analyses were conducted over 8 week follow-up; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.12 to 0.10]

2. Primary Outcome: Clinical Global Impression Scale - Severity (CGI-S)
Description: Clinical Global Impression Scale - Severity (CGI-S) is a 7-point scale is a clinician-completed measure that requires the clinician to rate the severity of the patient's illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of illness at the time of rating, with values ranging from 1 (normal, not at all ill), 2 (borderline ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), to 7 (extremely ill).
Time Frame: Weeks 0, 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  CGI-S Week 0 | 4.31 [3.93 to 4.69] | 4.39 [4.14 to 4.64]
  CGI-S Week 2 | 3.83 [3.45 to 4.21] | 4.03 [3.70 to 4.35]
  CGI-S Week 4 | 3.56 [3.25 to 3.87] | 3.86 [3.54 to 4.19]
  CGI-S Week 8 | 2.76 [2.38 to 3.13] | 3.51 [3.07 to 3.96]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.034, Chi-squared; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.15 to -0.01]

3. Primary Outcome: Abdominal Pain Index (API)
Description: The API is a well-validated and reliable measure of abdominal pain assessing the frequency, duration, and intensity of abdominal pain consisting of five items assessing the frequency, duration, and intensity of abdominal pain experienced during the prior 2 weeks. Two of the items are scored from 0 to 5, one is scaled 0 to 8, and two are scaled 0 to 10, with lower scores considered to be better than higher scores. Item scores are standardized using Z-scores and then summed to yield an index of abdominal pain that has been sensitive to change in previous epidemiological and treatment studies of FAP. Alpha reliability ranged from 0.80 to 0.93. The API will be a continuous primary outcome measure of abdominal pain.
Time Frame: Weeks 0, 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
score on a scale
  API-C Week 0 | 0.45 [0.20 to 0.69] | 0.47 [0.27 to 0.68]
  API-C Week 2 | -0.14 [-0.43 to 0.14] | 0.06 [-0.19 to 0.31]
  API-C Week 4 | -0.21 [-0.50 to 0.08] | 0.08 [-0.20 to 0.36]
  API-C Week 8 | -0.36 [-0.65 to -0.06] | -0.03 [-0.34 to 0.27]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.261, t-test, 2 sided; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.02]

4. Secondary Outcome: Pediatric Anxiety Rating Scale (PARS)
Description: Pediatric Anxiety Rating Scale (PARS) is a clinician administered measure of anxiety in children and adolescents. The PARS is comprised of a 50-item symptom checklist used to determine the presence or absence of specific anxiety symptoms during the prior week and 7 severity/impairment items, each scored from 0 to 5 . The the score on the 7 items allows the clinician to rate symptom severity and associated impairment on a range from 0 to 35, with higher scores reflecting greater symptom severity and associated impairment. The PARS is characterized by high interrater reliability (ICC = 0.97), adequate internal consistency (α = 0.64), and fair test-retest reliability (ICC = 0.55). There is preliminary support for convergent and divergent validity, and the PARS has demonstrated sensitivity to treatment effects in previously conducted clinical trials.
Time Frame: Weeks 0, 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  PARS Week 0 | 7.38 [5.66 to 9.11] | 9.73 [7.76 to 11.70]
  PARS Week 2 | 4.00 [2.81 to 5.19] | 6.78 [4.80 to 8.75]
  PARS Week 4 | 2.57 [1.55 to 3.59] | 5.76 [3.79 to 7.72]
  PARS Week 8 | 2.69 [1.66 to 3.73] | 5.55 [3.71 to 7.39]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.519, t-test, 2 sided; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.36 to 0.18]

5. Secondary Outcome: Children's Depression Rating Scale - Revised (CDRS-R)
Description: Children's Depression Rating Scale - Revised (CDRS-R) is a clinician administered measure of depression in children and adolescents and provides data necessary to diagnose depressive disorder and rate the severity of depressive symptoms over time. The CDRS-R is composed of 17 items, most rated on a 1 to 7 scale, with a minimum score of 17 and a maximum of 113. Higher scores reflect greater depression severity, with scores of 40 and above generally considered to be reflective of a depressive diagnosis.
Time Frame: Weeks 0, 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  CDRS-R Week 0 | 34.50 [30.32 to 38.68] | 39.23 [35.02 to 43.44]
  CDRS-R Week 2 | 27.81 [24.76 to 30.86] | 31.89 [27.80 to 35.99]
  CDRS-R Week 4 | 24.97 [22.31 to 27.62] | 28.35 [25.01 to 31.69]
  CDRS-R Week 8 | 23.88 [21.17 to 26.60] | 28.39 [23.32 to 33.47]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.704, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.77 to 0.52]

6. Secondary Outcome: Children's Global Assessment Scale (C-GAS)
Description: Children's Global Assessment Scale (C-GAS) is an interview-based adaptation of the Global Assessment Scale developed to assess child and adolescent functioning during a specified time period. Scores range from one to 100, with scores of 70 or below reflecting abnormally low functioning and higher scores reflecting better functioning. The C-GAS has demonstrated reliability, as well as discriminant and concurrent validity. A CGAS score of < 70 will be a requirement at study entry.
Time Frame: Weeks 0, 2, 4, and 8
Population: Analysis week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 40 | 41
units on a scale
  CGAS Week 0 | 54.42 [51.95 to 56.89] | 54.07 [51.77 to 56.38]
  CGAS Week 2 | 59.24 [55.98 to 62.49] | 58.05 [54.61 to 61.49]
  CGAS Week 4 | 63.27 [60.05 to 66.50] | 59.14 [56.10 to 62.17]
  CGAS Week 8 | 66.72 [62.74 to 70.70] | 61.22 [57.47 to 64.97]
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.046, t-test, 2 sided; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.01 to 1.17]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 31/40 | 36/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Citalopram (N=40) | Placebo (N=41)
gastric distress (Gastrointestinal disorders) | 13 | 14
appetite or weight change (Metabolism and nutrition disorders) | 11 | 20
vision disturbance (Eye disorders) | 2 | 3
dizziness (Nervous system disorders) | 16 | 16
headache (Nervous system disorders) | 31 | 36
itching (Skin and subcutaneous tissue disorders) | 11 | 8
fatigue (General disorders) | 20 | 28
nausea or vomiting (Gastrointestinal disorders) | 21 | 24
body aches (General disorders) | 29 | 31
palpitations (Cardiac disorders) | 12 | 12
bowel movement disturbance (Gastrointestinal disorders) | 20 | 21
eye irritation (Eye disorders) | 3 | 2
dry mouth (General disorders) | 5 | 2
earache (Ear and labyrinth disorders) | 5 | 4
nosebleed (General disorders) | 4 | 4
hearing disturbance (Ear and labyrinth disorders) | 5 | 4
throat pain (General disorders) | 11 | 10
motor disturbances (tics, twitches) (Nervous system disorders) | 5 | 3
urinary disturbance (Renal and urinary disorders) | 7 | 10
upper respiratory infection (Infections and infestations) | 10 | 11
sweating (General disorders) | 2 | 2
accidental injuries (General disorders) | 3 | 2
hyperactive (Nervous system disorders) | 11 | 18
aggression (Psychiatric disorders) | 3 | 1
nightmares (Psychiatric disorders) | 4 | 1
irritability (Psychiatric disorders) | 8 | 17
sleep disturbance (General disorders) | 21 | 28
anxiety and panic (Psychiatric disorders) | 7 | 15
mood lability (Psychiatric disorders) | 3 | 2
sadness, depression (Psychiatric disorders) | 9 | 10
memory disturbance (Nervous system disorders) | 3 | 1
fever (General disorders) | 2 | 2
hair loss (General disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Relatively small sample size, potentially without sufficient power to detect meaningful between group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No